CLINICAL TRIAL: NCT01243775
Title: Phase II Trial of First Line Docetaxel and Oxaliplatin in Stage IV or Relapsed Non-Small Cell Lung Cancer
Brief Title: BELotaxel(Docetaxel) and bellOXa(Oxaliplatin) in Advanced NSCLC
Acronym: BELOXAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: m601NSC10B
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belotaxel plus Belloxa (Experimental): Belotaxel 60 mg/m2 3 weekly (day 1) Belloxa 70 mg/m2 3 weekly (day 2)
  Interventions: Drug: Belotaxel; Drug: Belloxa

INTERVENTIONS:
Drug: Belotaxel — 60 mg/m2 3 weekly (day 1)
  Other Names: Docetaxel
Drug: Belloxa — 70 mg/m2 3 weekly (day 2)
  Other Names: Oxaliplatin

SUMMARY:
Lung cancer is the leading cause of cancer death in Korea as well as in other countries. About 80% of lung cancer is non-small cell lung cancer(NSCLC). The majority of patients with NSCLC require cytotoxic chemotherapy in the course of their illness. Combination chemotherapy using third generation anticancer drugs (paclitaxel, docetaxel, gemcitabine) with platinums(cisplatin or carboplatin) reached a plateau in their efficacy. Oxaliplatin, another platinum being used for colorectal, gastric and pancreatic cancer has lower adverse effects such as nausea and nephrotoxicity. In this phase II trial, we will observe efficacy and safety of docetaxel and oxaliplatin for patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB/IV or Relapsed NSCLC
* Age >= 18 years
* At least one measurable lesion by RECIST (version 1.1)
* ECOG PS 0, 1, 2
* Hematologic profile

  * Hgb > 8 g/dL, ANC >= 2,000/m3, Platelet >= 100,000/m3
* Hepatic profile

  * Total bilirubin <= 1.5 x upper normal value
  * Transaminases <= 3 x upper normal value <= 5 x upper normal value in case of liver metastasis
* Creatinine <= 1.5mg/dL
* Patients should be recovered from toxicities of previous treatment.
* Written informed consent by patient or surrogates

Exclusion Criteria:

* Patients who had been previously treated with chemotherapy for NSCLC
* Active infection requiring antibiotics treatment
* Prior diagnosis of other malignancy except radically treated basal cell or squamous cell carcinoma of the skin and carcinoma in situ of the uterine cervix
* Peripheral neuropathy >= grade 2 by NCI CTCAE 4.0
* Uncontrolled hypertension, Acute myocardial infarction within 6 months Unstable angina, Congestive heart failure >= NYHA grade 2 Uncontrolled significant arrhythmia
* Patients who entered other clinical trials within 4 weeks
* Pregnant or lactating women. women with child bearing age who are not willing to a contraceptive measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

REFERENCES:
- [Result] Ban H, Kim KS, Oh IJ, Yoon SH, Lee B, Yu J, Kim S, Lee HS, Shin HJ, Park CK, Kwon YS, Kim YI, Lim SC, Kim YC. Efficacy and safety of docetaxel plus oxaliplatin as a first-line chemotherapy in patients with advanced or metastatic non-small cell lung cancer. Thorac Cancer. 2014 Nov;5(6):525-9. doi: 10.1111/1759-7714.12123. Epub 2014 Oct 23. PMID 26767047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Belotaxel Plus Belloxa
Started | 33
Completed | 31
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Belotaxel Plus Belloxa
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Korean | 33
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 33

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: RECIST version 1.1
Time Frame: 6th week
Population: Intention to treat population
Measure: Number; unit: participants
Groups:
- Belotaxel Plus Belloxa: Belotaxel 60 mg/m2 3 weekly (day 1) plus Belloxa 70 mg/m2 3 weekly (day 2)
Arm/Group | Belotaxel Plus Belloxa
Number analyzed (Participants) | 33
participants | 11

2. Secondary Outcome: Progression Free Survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belotaxel Plus Belloxa
Number analyzed (Participants) | 33
months | 3.6 [2.8 to 4.5]

3. Secondary Outcome: Overall Survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belotaxel Plus Belloxa
Number analyzed (Participants) | 33
months | 10.9 [8.2 to 13.6]

4. Secondary Outcome: Neutropenia Grade 3-4
Description: Toxicity (CECAE ver 4.0) and Safety
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Belotaxel Plus Belloxa
Number analyzed (Participants) | 33
participants | 17

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Belotaxel Plus Belloxa
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belotaxel Plus Belloxa (N=33)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thromboembolism (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belotaxel Plus Belloxa (N=33)
Anorexia (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No